CLINICAL TRIAL: NCT02338284
Title: Optic Nerve Sheath Diameter Measured by Bedside Ultrasound May be a Simple Screening Test for Increased Intracranial Pressure in the Comatose Critically Ill Patient
Brief Title: Optic Nerve Sheath Diameter as a Screening Test for Increased Intracranial Pressure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Nawal Salahuddin, Consultant Physician, King Faisal Specialist Hospital & Research Center
Other Study IDs: 2141 103
Record Dates: First submitted 2015-01-06; First posted 2015-01-14 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Coma
Keywords: increased intracranial pressure; optic nerve sheath diameter
MeSH Terms: conditions — Coma; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: ultrasound of globe — * A high resolution 7.5 -10 MHz linear array ultrasound transducer probe will be used. A large amount of standard water-soluble ultrasound transmission gel will be applied to the patient's closed eyelid. The globe will be scanned in the transverse plane.• The ONSD will be measured at a predefined point 3 mm posterior to the globe in both eyes. • Measurement of the ONSD for both eyes will be done and the average the two measurements will be taken.
  * A value > 58mm (from reference 1) will be considered as indicative of increased ICP and the primary ICU team will be informed for rapid measures to decrease ICP or urgent imaging of the CNS.

SUMMARY:
Patients admitted to the ICU may have delayed awakening after their critical illness has resolved. Though most either are due to metabolic causes or delayed elimination of sedative medications, more serious pathologies such as intracranial hemorrhage, ischemic stroke, and vasogenic edema may also be the cause of coma. These pathologies all result in increases in intracranial pressure (ICP) with cerebral edema. Identifying elevated intracranial pressure elevations have so far, relied on invasive monitoring techniques requiring placement of an intracranial or intraventricular catheter.

The optic nerve sheath diameter (ONSD) has been described as a highly sensitive (88-94%) and specific (85% - 94%) noninvasive technique of identifying increased intracranial pressures in patients with brain trauma, intracranial bleeding or stroke[1-4]. This method requires placement of an ultrasound probe on the patient's closed eyelid and then a direct measurement of the diameter of the optic nerve sheath at a pre-specified distance from the globe. A value greater than 58 mm has been shown to correlate significantly with an increased ICP (> 20 cm H20); r = 0.71, p<0.001 [5].

The investigators hypothesize that bedside ultrasound measurement of the ONSD is a simple screening test for increased intracranial pressure and can be used to rapidly and efficiently identify patients in the ICU who have coma due to an increase in intracranial pressure. The investigators propose to carry out an observational trial to determine the predictive ability of the Optic Nerve Sheath Diameter for cerebral edema/ increased intracranial pressure and to compare it with the results of neuroimaging (CT and/or MRI).

DETAILED DESCRIPTION:
Patients admitted to the ICU may have delayed awakening after their critical illness has resolved. Though most either are due to metabolic causes or delayed elimination of sedative medications, more serious pathologies such as intracranial hemorrhage, ischemic stroke, and vasogenic edema may also be the cause of coma. These pathologies all result in increases in intracranial pressure (ICP) with cerebral edema. At this stage, the usual workup includes brain CT scans, MRI or EEG. These tests require transporting the patient from the ICU to the Radiology department, a process that may not be possible for an unstable, critically ill patient. Identifying elevated intracranial pressure elevations have so far, relied on invasive monitoring techniques requiring placement of an intracranial or intraventricular catheter.

The optic nerve attaches to the globe posteriorly and is wrapped in a sheath that contains cerebrospinal fluid. The optic nerve sheath is contiguous with the dura mater and has a trabeculated arachnoid space through which cerebrospinal fluid slowly percolates. Pressure increases around the brain are therefore transmitted to around the optic nerve and increase the diameter of the optic nerve sheath. This optic nerve sheath diameter (ONSD) has been described as a highly sensitive (88-94%) and specific (85% - 94%) noninvasive technique of identifying increased intracranial pressures in patients with brain trauma, intracranial bleeding or stroke[1-4]. This method requires placement of an ultrasound probe on the patient's closed eyelid and then a direct measurement of the diameter of the optic nerve sheath at a pre-specified distance from the globe. A value greater than 58 mm has been shown to correlate significantly with an increased ICP (> 20 cm H20); r = 0.71, p<0.001 [5].

We hypothesize that bedside ultrasound measurement of the ONSD is a simple screening test for increased intracranial pressure and can be used to rapidly and efficiently identify patients in the ICU who have coma due to an increase in intracranial pressure.

Objectives:

To determine the role of bedside ONSD measurement by ultrasound in the evaluation of comatose patients in the ICU.

METHODS:

* Study Design: Prospective, Observational study
* Study Sample:

  * Inclusion criteria: Consecutive, adult patients already admitted to the critical care service and in whom a cause of coma is not determined.
  * Exclusion criteria: obvious ocular trauma, patients on sedative or narcotic infusions.

Variables to be measured:

Independent variables:

Demographic identifiers; age, gender, comorbidity, admitting diagnosis, APACHE II scores, SAPS II scores

Dependent (Outcome) variables:

1. Diagnosis of cerebral edema/ elevated intracranial pressure as measured by Optic nerve sheath diameter
2. Diagnosis of cerebral edema/ elevated intracranial pressure as measured by neuroimaging
3. ICU mortality

Materials & Methodologies:

1. Screening & Enrollment of patients:

   1. All ICU patients will be screened for enrollment.
   2. For patients meeting the inclusion criteria, informed consent will be obtained from the patient or family members at bedside.
   3. Demographic information will be collected in Case Record Forms (Appendix 2: Sample CRF)
   4. Ultrasound examinations will be carried out and results entered into a CRF.
2. Technique of ONSD ultrasound measurement from Reference 6.

   * A high resolution 7.5 -10 MHz linear array ultrasound transducer probe will be used. A large amount of standard water-soluble ultrasound transmission gel will be applied to the patient's closed eyelid. The globe will be scanned in the transverse plane.
   * The ONSD will be measured at a predefined point 3 mm posterior to the globe in both eyes.
   * Measurement of the ONSD for both eyes will be done and the average the two measurements will be taken.
   * A value > 58mm (from reference 1) will be considered as indicative of increased ICP and the primary ICU team will be informed for rapid measures to decrease ICP or urgent imaging of the CNS.
3. Statistical Methods:

   1. Sample size & Sampling: Consecutive admissions to the ICU will be enrolled. Since this is a proof of concept study, the projected sample size is 40 patients. An interim analysis will be carried out after 20 patients are enrolled and a further 20 will be enrolled as necessary
   2. Analysis: Categorical variables will be reported as proportions or percentages, continuous variables as means or medians. Differences between groups will be estimated using CHI2, student t test or Mann-Whitney U test, as appropriate. A p value =0.05 will be considered significant. SPSS version 22.0 will be used for all analysis.

Ethical considerations:

* Informed Consent for ultrasonographic examination. The use of use of ultrasound for the assessment and management of critically ill patients in the ICU and emergency room is considered as standard of care and is routinely practiced in ICUs around the world. Since ultrasound evaluation has become incorporated into usual ICU practice, written consent is not required in its routine use. We therefore ask for a waiver of informed consent since we will not be performing any deviation from usual ICU care and our study is simply a collection of practice into a protocolized form.
* Research Advisory Committee (RAC) Review This protocol will be reviewed and approved by the hospital Research Advisory committee responsible for oversight of the study.

  2. Subject Confidentiality & Protection of Rights of Control Subjects All case record forms, reports and other records will be identified only by the Study Identification Number (SID) to maintain subject confidentiality. All records will be kept in a password-protected file. All computer entry and networking programs will be done using SIDs only.

  3. Study Modification/Discontinuation The study may be modified or discontinued at any time by the primary investigators and or Research Advisory Committee as part of their duties to ensure that research subjects are protected.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive, adult patients already admitted to the critical care service and in whom a cause of coma is not determined.

Exclusion Criteria:

* Obvious ocular trauma
* Patients on sedative or narcotic infusions

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive, adult patients already admitted to the critical care service with unexplained coma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Cerebral edema by Optic nerve sheath diameter | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: nawal salahuddin, MD,FCCP, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal Specialist Hospital & Research Centre, Riyadh, Ar-Riyadh, Saudi Arabia